CLINICAL TRIAL: NCT04398706
Title: Safety and Immunogenicity of a Pneumococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Toddlers and Infants
Brief Title: Study of a Pneumococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Toddlers and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK00008; U1111-1238-1638 (Registry Identifier: ICTRP); PSK00008 (Other: Sanofi Identifier)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Immunisation; Diphtheria Immunisation; Tetanus Immunisation; Pertussis Immunisation; Hepatitis B Immunisation; Haemophilus Influenzae Type b Immunisation; Polio Immunisation; Measles Immunisation; Rubella Immunisation; Varicella Immunisation; Mumps Immunisation
MeSH Terms: interventions — Herpes Zoster Vaccine; Chickenpox Vaccine; Measles-Mumps-Rubella Vaccine; 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin); Tetanus Toxoid; pentacel; Rotavirus Vaccines; RotaTeq; Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a modified double-blind fashion:
  * Investigators and study staff who conduct the safety assessment and the participant will not know which vaccine is administered
  * Only the study staff who prepare and administer the vaccine and are not involved with the safety evaluation will know which vaccine is administered This study will be observer-blinded between any SP0202 formulation and Prevnar 13 and double-blind across the 3 SP0202 formulations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Group 1 (Experimental): One dose of SP0202-IIb and one dose of DTaP-IPV// Hib vaccine in toddlers aged 12-15 months who have previously received the 3-dose primary series of Prevnar13
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 1; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate)
- Group 2 (Experimental): One dose of SP0202-VI and one dose of DTaP-IPV// Hib vaccine in toddlers aged 12-15 months who have previously received the 3-dose primary series of Prevnar13
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 2; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate)
- Group 3 (Experimental): One dose of SP0202-VII and one dose of DTaP-IPV// Hib vaccine in toddlers aged 12-15 months who have previously received the 3-dose primary series of Prevnar13
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 3; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate)
- Group 4 (Active Comparator): One dose of Prevnar 13 and one dose of DTaP-IPV// Hib vaccine in toddlers aged 12-15 months who have previously received the 3-dose primary series of Prevnar13
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate)
- Group 5 (Experimental): Four doses of SP0202-IIb at 2, 4, 6 and 12-15 months Routine pediatric vaccines: DTaP-IPV// Hib vaccine, rotavirus vaccine at 2, 4, 6 months; MMR vaccine and varicella vaccine at 12-15 months Hepatitis B vaccine at 2, 4, 6 months, as applicable
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 1; Biological: Varicella Virus Vaccine Live; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate); Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine* [Recombinant] *as applicable
- Group 6 (Experimental): Four doses of SP0202-VI at 2, 4, 6 and 12-15 months Routine pediatric vaccines: DTaP-IPV// Hib vaccine, rotavirus vaccine at 2, 4, 6 months; MMR vaccine and varicella vaccine at 12-15 months Hepatitis B vaccine at 2, 4, 6 months, as applicable
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 2; Biological: Varicella Virus Vaccine Live; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate); Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine* [Recombinant] *as applicable
- Group 7 (Experimental): Four doses of SP0202-VII at 2, 4, 6 and 12-15 months Routine pediatric vaccines: DTaP-IPV// Hib vaccine, rotavirus vaccine at 2, 4, 6 months; MMR vaccine and varicella vaccine at 12-15 months Hepatitis B vaccine at 2, 4, 6 months, as applicable
  Interventions: Biological: Pneumococcal Conjugate Vaccine formulation 3; Biological: Varicella Virus Vaccine Live; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate); Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine* [Recombinant] *as applicable
- Group 8 (Active Comparator): Four doses of Prevnar 13 at 2, 4, 6 and 12-15 months Routine pediatric vaccines: DTaP-IPV// Hib vaccine, rotavirus vaccine at 2, 4, 6 months; MMR vaccine and varicella vaccine at 12-15 months Hepatitis B vaccine at 2, 4, 6 months, as applicable
  Interventions: Biological: Varicella Virus Vaccine Live; Biological: Measles, Mumps, and Rubella Virus Vaccine Live; Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]; Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate); Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Hepatitis B Vaccine* [Recombinant] *as applicable

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine formulation 1 — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: SP0202-IIb
  Arms: Group 1; Group 5
Biological: Pneumococcal Conjugate Vaccine formulation 2 — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: SP0202-VI
  Arms: Group 2; Group 6
Biological: Pneumococcal Conjugate Vaccine formulation 3 — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: SP0202-VII
  Arms: Group 3; Group 7
Biological: Varicella Virus Vaccine Live — Pharmaceutical form:liquid Route of administration: subcutaneous
  Other Names: Varicella vaccine, VARIVAX®
  Arms: Group 5; Group 6; Group 7; Group 8
Biological: Measles, Mumps, and Rubella Virus Vaccine Live — Pharmaceutical form:liquid Route of administration: subcutaneous
  Other Names: MMR vaccine, M-M-R ®II
  Arms: Group 5; Group 6; Group 7; Group 8
Biological: Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein] — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: Prevnar 13®
  Arms: Group 4; Group 8
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate) — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: DTaP-IPV// Hib vaccine, Pentacel®
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Pharmaceutical form:liquid Route of administration: oral
  Other Names: Rotavirus vaccine, RotaTeq
  Arms: Group 5; Group 6; Group 7; Group 8
Biological: Hepatitis B Vaccine* [Recombinant] *as applicable — Pharmaceutical form:liquid Route of administration: intramuscular
  Other Names: Hepatitis B vaccine, ENGERIX-B®
  Arms: Group 5; Group 6; Group 7; Group 8

SUMMARY:
Primary objectives:

* To assess the safety profile of each SP0202 formulation and Prevnar 13 in toddlers and infants (after each and any injection).
* To assess the immune response (serotype specific IgG concentration) of the SP0202 formulations and Prevnar 13 1 month after the administration of one dose in toddlers (Groups 1-4)
* To assess the immune response (serotype specific IgG concentration) of the SP0202 formulations and Prevnar 13 1 month after the administration of 3 doses in infants (Groups 5-8)
* To assess the immune response (serotype specific IgG concentration) of the SP0202 formulations and Prevnar 13 1 month after administration of a 4-dose schedule in infants (Groups 5-8)

Secondary objectives:

* To assess the immune response (serotype specific OPA titer) of the SP0202 formulations and Prevnar 13 1 month after the administration of one dose in toddlers (Groups 1-4)
* To assess the immune response (serotype specific OPA titer) of the SP0202 formulations and Prevnar 13 1 month after the administration of 3 doses in a subset of infants (Groups 5-8)
* To assess the immune response (serotype specific OPA titer) of the SP0202 formulations and Prevnar 13 1 month after administration of a 4-dose schedule in a subset of infants (Groups 5-8)
* In toddlers: to describe the Ab responses against Pentacel antigens before and 1 month following injection of Pentacel
* In infants: to describe the Ab responses against antigens of the routine pediatric vaccines (Pentacel, RotaTeq, ENGERIX-B, M-M-RII, and VARIVAX) when administered concomitantly with either SP0202 or Prevnar 13 (at pre-Dose 1 (as applicable) for RotaTeq, Diphteria, Tetanus and Pertussis antigens; at PD3 for ENGERIX-B, RotaTeq, and Pentacel; at PD4 for M-M-RII and VARIVAX])

DETAILED DESCRIPTION:
For toddlers, the duration of each participant's participation in the study will be approximately 6 months for subjects enrolled in Groups 1, 2, 3, and 4.

For infants, the duration of each participant's participation in the study will be approximately 16 to 19 months for subjects enrolled in Groups 5, 6, 7, and 8.

ELIGIBILITY:
Inclusion criteria :

Toddlers and infants:

* Participant and parent/guardian are able to attend all scheduled visits and to comply with all study procedures
* Born at full term of pregnancy (≥ 37 weeks) and/or with a birth weight ≥ 5.5 lbs or 2.5 kg

Specifically for toddlers:

* Aged 12 to 15 months on the day of the first study visit
* Participant has received 3 doses of Prevnar 13 and 3 doses of diphteria, tetanus, acellular pertussis, poliovirus and Haemophilus influenzae type b antigens in infancy

Specifically for infants:

- Aged 42 to 89 days on the day of the first study visit

Exclusion criteria:

Toddlers and infants

* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated
* Blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
* Active tuberculosis
* History of S. pneumoniae infection or disease, confirmed either serologically or microbiologically
* History of any neurologic disorder, including any seizures and progressive neurologic disorders
* History of Guillain-Barré syndrome
* Known systemic hypersensitivity to any of the vaccine components or to latex, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Verbal report of thrombocytopenia contraindicating intramuscular vaccination in the Investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Chronic illness (including, but not limited to, cardiac disorders, congenital heart disease, chronic lung disease, renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and know congenital or genetic diseases) that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives
* In an emergency setting, or hospitalized involuntarily
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C / ≥ 100.4 F). A prospective participant should not be included in the study until the condition has resolved or until 3 days after the febrile event has resolved
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study Specifically for toddlers
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine from enrollment through the last blood sampling Visit (Visit 2), except for influenza vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of diphtheria, tetanus, pertussis, poliomyelitis, and/or H. influenzae type b infection or disease Specifically for infants
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine from enrollment through the last blood sampling Visit (Visit 6), except for influenza vaccination or COVID-19 vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines, and COVID-19 vaccines as applicable per local recommendations
* Receipt of immune globulins, blood or blood-derived products since birth.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth
* Previous vaccination against S. pneumoniae
* Previous vaccination against the following antigens: diphteria, tetanus, pertussis, H. influenzae type b, poliovirus, rotavirus, measles, mumps, rubella, and varicella
* Receipt of more than 1 previous dose of hepatitis B vaccine
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, measles, mumps, rubella, varicella, H. influenzae type b, and/or rotavirus infection or disease
* History of intussusception

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 42 Days to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 852 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (57):
- United States (49):
  - The Children's Clinic Of Jonesboro PA Site Number : 8400143, Jonesboro, Arkansas
  - Southland Clinical Research Center Site Number : 8400040, Bellflower, California
  - Joint Clinical Trials Huntington Park Site Number : 8400030, Huntington Park, California
  - Matrix Clinical Research Huntington Park Site Number : 8400058, Huntington Park, California
  - Matrix Clinical Research Site Number : 8400059, Los Angeles, California
  - Orange County Research Institute Site Number : 8400060, Ontario, California
  - California Research Foundation Site Number : 8400052, San Diego, California
  - Meridian Clinical Research Washington DC Site Number : 8400119, Washington D.C., District of Columbia
  - International Research Partners, LLC Site Number : 8400077, Doral, Florida
  - Homestead Medical Clinic, P.A. Site Number : 8400032, Homestead, Florida
  - Dade Research Center Site Number : 8400122, Miami, Florida
  - Miami Clinical Research Site Number : 8400020, Miami, Florida
  - Amber Clinical Research, LLC Site Number : 8400019, Miami, Florida
  - Jedidiah Clinical Research Site Number : 8400049, Tampa, Florida
  - Javara Albany Site Number : 8400140, Albany, Georgia
  - Centricity Research Talbotton - DBA IACT Health Research at Talbotton Site Number : 8400062, Columbus, Georgia
  - Javara Fayetteville Site Number : 8400139, Fayetteville, Georgia
  - Dumog Research Site Number : 8400134, Smyrna, Georgia
  - Bingham Memorial Hospital Site Number : 8400067, Blackfoot, Idaho
  - Leavitt Clinical Research Site Number : 8400127, Idaho Falls, Idaho
  - Hutchinson Clinic Site Number : 8400074, Hutchinson, Kansas
  - Qualmedica Research, LLC Site Number : 8400084, Bowling Green, Kentucky
  - Michael W. Simon, MD, PSC Site Number : 8400002, Lexington, Kentucky
  - Meridian Clinical Research, LLC Site Number : 8400112, Baton Rouge, Louisiana
  - Benchmark Research Site Number : 8400012, Covington, Louisiana
  - Velocity Clinical Research Lafayette Site Number : 8400132, Lafayette, Louisiana
  - Javara Annapolis Site Number : 8400137, Annapolis, Maryland
  - Javara Chevy Chase Site Number : 8400138, Chevy Chase, Maryland
  - Children's Mercy Hospital Site Number : 8400008, Kansas City, Missouri
  - Boeson Research Site Number : 8400004, Missoula, Montana
  - Meridian Clinical Research Site Number : 8400102, Grand Island, Nebraska
  - Lincoln Pediatric Group Site Number : 8400125, Lincoln, Nebraska
  - Pediatric Infectious Diseases Research Site Number : 8400104, Omaha, Nebraska
  - Atrium Health Site Number : 8400124, Charlotte, North Carolina
  - Ardmore Medical Research Site Number : 8400043, Winston-Salem, North Carolina
  - Pediatric Associates of Mt. Carmel Site Number : 8400005, Cincinnati, Ohio
  - Cheraw Pediatrics Site Number : 8400017, Cheraw, South Carolina
  - Tribe Clinical Research Site Number : 8400025, Greenville, South Carolina
  - Javara Dallas Site Number : 8400135, Dallas, Texas
  - Pininos Pediatric Services Site Number : 8400121, El Paso, Texas
  - North Texas Clinical Trials Site Number : 8400015, Fort Worth, Texas
  - Houston Clinical Research Associates Site Number : 8400023, Houston, Texas
  - FMC Science, LLC Site Number : 8400086, Lampasas, Texas
  - DCOL Center for Clinical Research Site Number : 8400107, Longview, Texas
  - Biopharma Informatic Site Number : 8400066, McAllen, Texas
  - Benchmark Research San Antonio Site Number : 8400129, San Antonio, Texas
  - Sun Research Institute Site Number : 8400011, San Antonio, Texas
  - Tekton Research Site Number : 8400076, San Antonio, Texas
  - MultiCare Institute for Research & Innovation Site Number : 8400024, Spokane, Washington
- Canada (3):
  - Investigational Site Number : 1240002, Vancouver, British Columbia
  - Investigational Site Number : 1240001, Halifax, Nova Scotia
  - Investigational Site Number : 1240006, Hamilton, Ontario
- Honduras (2):
  - Investigational Site Number : 3400002, Municipio Del Distrito Central
  - Investigational Site Number : 3400001, San Pedro Sula
- Puerto Rico (3):
  - Investigational Site Number : 6300002, Bayamón
  - Investigational Site Number : 6300004, Guayama
  - Investigational Site Number : 6300001, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PSK00008 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25336&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Stage I of study was conducted at 22 active centers in the US between 22 May 2020 and 10 March 2021. The Stage II of study was conducted at 35 active centers in the US, Canada and Honduras between 16 April 2021 and 24 February 2022.
Pre-assignment Details: A total of 140 participants were randomized in Stage I and 712 participants were randomized in Stage II of study.
Groups:
- Stage I: Group 1 SP0202-IIb: Toddlers aged between 12 and 15 months who previously received the 3-dose primary series of Prevnar 13 received 1 dose of SP0202-IIb formulation, concomitantly administered with Pentacel.
- Stage I: Group 2 SP0202-VI: Toddlers aged between 12 and 15 months who previously received the 3-dose primary series of Prevnar 13 received 1 dose of SP0202-VI formulation, concomitantly administered with Pentacel.
- Stage I: Group 3 SP0202-VII: Toddlers aged between 12 and 15 months who previously received the 3-dose primary series of Prevnar 13 received 1 dose of SP0202-VII formulation, concomitantly administered with Pentacel.
- Stage I: Group 4 Prevnar 13: Toddlers aged between 12 and 15 months who previously received the 3-dose primary series of Prevnar 13 received another dose of Prevnar 13, concomitantly administered with Pentacel.
- Stage II: Group 5 SP0202-IIb: Infants aged 2 months received 3 doses of SP0202-IIb formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age [that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII (measles, mumps, and rubella) and Varivax at 12 to 15 months of age].
- Stage II: Group 6 SP0202-VI: Infants aged 2 months received 3 doses of SP0202-VI formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Stage II: Group 7 SP0202-VII: Infants aged 2 months received 3 doses of SP0202-VII formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Stage II: Group 8 Prevnar 13: Infants aged 2 months received 3 doses of Prevnar 13 at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
Period: Overall Study
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Started | 35 | 35 | 35 | 35 | 179 | 178 | 179 | 176
Completed | 35 | 31 | 32 | 32 | 148 | 147 | 151 | 160
Not Completed | 0 | 4 | 3 | 3 | 31 | 31 | 28 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1 | 6 | 3 | 8 | 2
Not completed — Withdrawal by parent/guardian | 0 | 2 | 1 | 2 | 19 | 23 | 13 | 11
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 6 | 4 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Stage II: Group 5 SP0202-IIb: Infants aged 2 months received 3 doses of SP0202-IIb formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Stage II: Group 6 SP0202-VI: Infants aged 2 months were received 3 doses of SP0202-VI formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Stage II: Group 7 SP0202-VII: Infants aged 2 months were received 3 doses of SP0202-VII formulation at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Stage II: Group 8 Prevnar 13: Infants aged 2 months were received 3 doses of Prevnar 13 at 2, 4, and 6 months of age and fourth dose at 12 to 15 months of age, co-administered with pediatric vaccines recommended at this age (that is, Pentacel, RotaTeq and Engerix-B at 2, 4 and 6 months of age and M-M-RII and Varivax at 12 to 15 months of age).
- Total: Total of all reporting groups
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13 | Total
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 179 | 178 | 179 | 176 | 852
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.1 (0.11) | 1.1 (0.10) | 1.1 (0.12) | 1.2 (0.11) | 0.2 (0.03) | 0.2 (0.03) | 0.2 (0.03) | 0.2 (0.03) | 0.3 (0.36)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17 | 12 | 20 | 17 | 93 | 94 | 78 | 90 | 421
  Male | 18 | 22 | 15 | 18 | 86 | 84 | 101 | 86 | 430
  Missing | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 2 | 26 | 26 | 23 | 23 | 103
  Asian | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 8
  Black or African American | 5 | 2 | 3 | 6 | 10 | 17 | 10 | 11 | 64
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 24 | 28 | 29 | 25 | 75 | 67 | 79 | 80 | 407
  Multiple | 2 | 3 | 0 | 0 | 64 | 67 | 67 | 59 | 262
  Not Reported | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4
  Unknown | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Missing | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant or in a clinical investigation participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. Immediate events were recorded to capture medically relevant unsolicited systemic AEs (including those related to the product administered) that occurred within the first 30 minutes after vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination and included both serious adverse events (SAEs) and non-serious unsolicited AEs.
Time Frame: Up to 30 minutes after each vaccination
Population: Analysis was performed on the Safety analysis set (SafAS) that included all participants who received at least 1 dose of the study vaccines and had any safety data available. One participant who was randomized to the reporting group "Stage II: Group 7 SP0202-VII" was administered SP0202-IIb formulation. Therefore, the participant was included in "Stage II: Group 5 SP0202-IIb" for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 35 | 34 | 35 | 34 | 180 | 178 | 176 | 176
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted in the protocol and CRB and were considered to be related to the product administered. An injection site reaction was an adverse reaction at and around the injection site which were commonly inflammatory reactions. Solicited injection site reactions included tenderness, erythema and swelling around the injection site and were planned to be collected and reported for SP0202/Prevnar 13 for both toddlers and infants.
Time Frame: Up to 7 days after each vaccination
Population: Analysis was performed on SafAS. One participant who was randomized to the reporting group "Stage II: Group 7 SP0202-VII" was administered SP0202-IIb formulation. Therefore, the participant was included in "Stage II: Group 5 SP0202-IIb" for analysis. Only participants with data collected for each specified category are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 31 | 32 | 31 | 30 | 168 | 170 | 168 | 171
Participants | 21 | 18 | 21 | 13 | 119 | 128 | 126 | 124

3. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB and considered as related to the product administered. Solicited systemic reactions included fever, vomiting, abnormal crying, drowsiness, appetite loss, and irritability. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Up to 7 days after each vaccination
Population: Analysis was performed on SafAS. One participant who was randomized to the reporting group "Stage II: Group 7 SP0202-VII" was administered SP0202-IIb formulation. Therefore, the participant was included in "Stage II: Group 5 SP0202-IIb" for analysis. Only participants with data collected for this outcome measure are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 33 | 33 | 33 | 30 | 168 | 169 | 168 | 171
Participants | 25 | 23 | 27 | 24 | 139 | 143 | 137 | 138

4. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product, and which did not necessarily have a causal relationship with this treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset window post-vaccination. Unsolicited AEs included both SAEs and non-serious unsolicited AEs. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Up to 30 days after each vaccination
Population: Analysis was performed on SafAS. One participant who was randomized to the reporting group "Stage II: Group 7 SP0202-VII" was administered SP0202-IIb formulation. Therefore, the participant was included in "Stage II: Group 5 SP0202-IIb" for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 35 | 34 | 35 | 34 | 180 | 178 | 176 | 176
Participants | 7 | 3 | 4 | 6 | 122 | 116 | 118 | 117

5. Primary Outcome: Number of Participants With SAEs and Adverse Event of Special Interest (AESIs)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. The following AE were captured as AESI throughout the study: Anaphylaxis defined as per the Brighton collaboration case definition, convulsions including febrile convulsions, hypotonic-hyporesponsive episode and apnea. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: From first dose vaccine administration (Day 1) until 6 months after the last dose administration, 490 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 35 | 34 | 35 | 34 | 180 | 178 | 176 | 176
Participants
  Any SAEs | 0 | 1 | 0 | 0 | 3 | 9 | 8 | 9
  Any AESIs | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0

6. Primary Outcome: For Toddlers: Serotype Specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for Each Pneumococcal Serotype at 30 Days Post-Dose
Description: The GMCs for serotype specific pneumococcal IgG antibodies were measured using pneumococcal capsular polysaccharide-electro-chemiluminescent assay (PnPS-ECL), a multiplexed serological assay which allows for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens.
Time Frame: Day 30
Population: Per protocol analysis set 1 (PPAS1) was a subset of Full analysis set (FAS)1. FAS1: All randomized participants to Groups 1 to 4 who received at least 1 dose of study vaccine and had a valid post vaccination blood sample result [serotype specific IgG concentration or serotype specific opsonophagocytic activity (OPA) titer for at least 1 serotype, or titer/concentration for at least 1 antigen on concomitant vaccines]. Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram/millilitre (mcg/mL)
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13
Number analyzed (Participants) | 25 | 26 | 27 | 29
microgram/millilitre (mcg/mL)
  Serotype 1 | 2.46 [1.59 to 3.82] | 2.12 [1.40 to 3.21] | 3.29 [2.55 to 4.24] | 3.80 [2.76 to 5.24]
  Serotype 3: number analyzed (Participants) | 25 | 26 | 27 | 28
  Serotype 3 | 0.766 [0.569 to 1.03] | 0.973 [0.748 to 1.26] | 1.16 [0.963 to 1.40] | 0.835 [0.629 to 1.11]
  Serotype 4 | 1.53 [1.07 to 2.19] | 1.51 [1.10 to 2.08] | 2.27 [1.58 to 3.27] | 1.73 [1.32 to 2.25]
  Serotype 5 | 2.44 [1.74 to 3.42] | 2.38 [1.66 to 3.42] | 2.80 [2.00 to 3.93] | 2.69 [2.02 to 3.58]
  Serotype 6A | 7.53 [5.48 to 10.4] | 5.87 [4.20 to 8.20] | 8.29 [6.51 to 10.6] | 8.54 [6.44 to 11.3]
  Serotype 6B | 5.21 [3.67 to 7.40] | 4.16 [3.15 to 5.50] | 7.11 [5.21 to 9.70] | 5.77 [4.33 to 7.70]
  Serotype 7F | 2.99 [2.32 to 3.86] | 3.23 [2.37 to 4.41] | 2.91 [2.23 to 3.80] | 3.80 [3.06 to 4.73]
  Serotype 9V: number analyzed (Participants) | 25 | 26 | 27 | 28
  Serotype 9V | 3.25 [2.47 to 4.27] | 2.99 [2.22 to 4.01] | 5.27 [3.99 to 6.97] | 3.13 [2.31 to 4.24]
  Serotype 14 | 7.37 [5.39 to 10.1] | 6.54 [4.62 to 9.27] | 5.75 [4.48 to 7.38] | 9.83 [7.65 to 12.6]
  Serotype 18C | 1.80 [1.25 to 2.59] | 2.23 [1.57 to 3.19] | 2.19 [1.67 to 2.87] | 2.53 [1.99 to 3.21]
  Serotype 19A | 3.67 [2.56 to 5.26] | 5.41 [3.62 to 8.08] | 5.45 [4.17 to 7.11] | 6.20 [4.83 to 7.96]
  Serotype 19F | 3.88 [2.77 to 5.42] | 4.12 [2.99 to 5.70] | 5.79 [4.02 to 8.35] | 6.50 [4.69 to 9.02]
  Serotype 23F | 2.42 [1.71 to 3.43] | 2.65 [1.98 to 3.55] | 3.64 [2.75 to 4.82] | 3.02 [2.11 to 4.32]
  Serotype 8 | 6.86 [4.96 to 9.50] | 4.91 [3.74 to 6.44] | 7.11 [5.17 to 9.80] | 0.235 [0.158 to 0.350]
  Serotype 9N | 3.46 [2.21 to 5.43] | 2.02 [1.43 to 2.84] | 2.78 [2.04 to 3.79] | 0.668 [0.437 to 1.02]
  Serotype 10A: number analyzed (Participants) | 25 | 26 | 27 | 27
  Serotype 10A | 1.84 [1.18 to 2.87] | 1.05 [0.669 to 1.66] | 1.48 [0.988 to 2.21] | 0.244 [0.180 to 0.331]
  Serotype 11A | 4.41 [3.25 to 5.99] | 3.20 [2.48 to 4.13] | 4.61 [3.34 to 6.35] | 0.188 [0.144 to 0.247]
  Serotype 12F: number analyzed (Participants) | 25 | 25 | 27 | 28
  Serotype 12F | 0.767 [0.454 to 1.29] | 0.778 [0.541 to 1.12] | 0.907 [0.596 to 1.38] | 0.094 [0.078 to 0.112]
  Serotype 15B | 0.680 [0.447 to 1.03] | 0.560 [0.370 to 0.848] | 0.644 [0.425 to 0.974] | 0.172 [0.122 to 0.241]
  Serotype 22F | 4.43 [3.12 to 6.30] | 4.26 [2.66 to 6.82] | 5.20 [3.51 to 7.69] | 0.178 [0.122 to 0.259]
  Serotype 33F: number analyzed (Participants) | 25 | 26 | 27 | 27
  Serotype 33F | 1.26 [0.694 to 2.29] | 1.13 [0.771 to 1.65] | 1.75 [1.09 to 2.79] | 0.256 [0.189 to 0.345]

7. Primary Outcome: For Infants: Percentage of Participants With Serotype Specific IgG Concentration >=0.35 mcg/mL 30 Days Post-Dose 3
Description: Percentage of infants with serotype specific IgG concentration >=0.35 mcg/mL for each pneumococcal serotype included in the SP0202 formulations were measured using ECL, a multiplexed serological assay which allows for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens.
Time Frame: Day 150
Population: Per protocol analysis set 2 (PPAS2) was a subset of FAS2. FAS2: All randomized participants to Groups 5 to 8 who received at least 1 dose of study vaccine in primary series and had a valid post-primary series vaccination blood sample result (serotype specific IgG concentration or serotype specific OPA titer for at least 1 serotype, or titer/concentration for at least 1 antigen on concomitant vaccines). Only participants with data collected for each specified category are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 133 | 122 | 125 | 132
percentage of participants
  Serotype 1 | 97.7 [93.5 to 99.5] | 96.7 [91.8 to 99.1] | 95.2 [89.8 to 98.2] | 97.0 [92.4 to 99.2]
  Serotype 3 | 94.7 [89.5 to 97.9] | 95.1 [89.6 to 98.2] | 97.6 [93.1 to 99.5] | 81.8 [74.2 to 88.0]
  Serotype 4 | 97.0 [92.5 to 99.2] | 95.9 [90.7 to 98.7] | 97.6 [93.1 to 99.5] | 97.7 [93.5 to 99.5]
  Serotype 5 | 98.5 [94.7 to 99.8] | 96.7 [91.8 to 99.1] | 93.6 [87.8 to 97.2] | 97.0 [92.4 to 99.2]
  Serotype 6A | 99.2 [95.9 to 100] | 96.7 [91.8 to 99.1] | 99.2 [95.6 to 100] | 99.2 [95.9 to 100]
  Serotype 6B | 85.7 [78.6 to 91.2] | 81.1 [73.1 to 87.7] | 84.0 [76.4 to 89.9] | 97.0 [92.4 to 99.2]
  Serotype 7F | 100 [97.3 to 100] | 100 [97.0 to 100] | 99.2 [95.6 to 100] | 100 [97.2 to 100]
  Serotype 9V | 96.2 [91.4 to 98.8] | 89.3 [82.5 to 94.2] | 94.4 [88.8 to 97.7] | 99.2 [95.9 to 100]
  Serotype 14: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 14 | 99.2 [95.9 to 100] | 99.2 [95.5 to 100] | 97.6 [93.1 to 99.5] | 96.9 [92.4 to 99.2]
  Serotype 18C | 97.0 [92.5 to 99.2] | 97.5 [93.0 to 99.5] | 97.6 [93.1 to 99.5] | 96.2 [91.4 to 98.8]
  Serotype 19A | 94.0 [88.5 to 97.4] | 93.4 [87.5 to 97.1] | 96.0 [90.9 to 98.7] | 97.0 [92.4 to 99.2]
  Serotype 19F: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 19F | 100 [97.3 to 100] | 99.2 [95.5 to 100] | 96.8 [92.0 to 99.1] | 99.2 [95.8 to 100]
  Serotype 23F | 97.7 [93.5 to 99.5] | 96.7 [91.8 to 99.1] | 96.0 [90.9 to 98.7] | 93.9 [88.4 to 97.3]
  Serotype 8: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 8 | 99.2 [95.9 to 100] | 100 [97.0 to 100] | 99.2 [95.6 to 100] | 9.2 [4.8 to 15.5]
  Serotype 9N | 99.2 [95.9 to 100] | 98.4 [94.2 to 99.8] | 98.4 [94.3 to 99.8] | 65.9 [57.2 to 73.9]
  Serotype 10A: number analyzed (Participants) | 133 | 122 | 120 | 132
  Serotype 10A | 93.2 [87.5 to 96.9] | 92.6 [86.5 to 96.6] | 96.0 [90.9 to 98.7] | 3.8 [1.2 to 8.6]
  Serotype 11A | 98.5 [94.7 to 99.8] | 100 [97.0 to 100] | 97.6 [93.1 to 99.5] | 7.6 [3.7 to 13.5]
  Serotype 12F | 97.7 [93.5 to 99.5] | 93.4 [87.5 to 97.1] | 94.4 [88.8 to 97.7] | 0 [0 to 2.8]
  Serotype 15B: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 15B | 98.5 [94.7 to 99.8] | 95.9 [90.7 to 98.7] | 97.6 [93.1 to 99.5] | 6.9 [3.2 to 12.6]
  Serotype 22F | 100 [97.3 to 100] | 97.5 [93.0 to 99.5] | 97.6 [93.1 to 99.5] | 3.0 [0.8 to 7.6]
  Serotype 33F: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 33F | 91.7 [85.7 to 95.8] | 89.3 [82.5 to 94.2] | 92.8 [86.8 to 96.7] | 3.8 [1.3 to 8.7]

8. Primary Outcome: For Infants: Serotype Specific IgG GMCs for Each Pneumococcal Serotype at 30 Days Post-Dose 3
Description: The GMCs for serotype-specific pneumococcal IgG antibodies were measured using PnPS-ECL, a multiplexed serological assay which allows for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens.
Time Frame: Day 150
Population: PPAS2 was a subset of FAS2. FAS2: All randomized participants to Groups 5 to 8 who received at least 1 dose of study vaccine in primary series and had a valid post-primary series vaccination blood sample result (serotype specific IgG concentration or serotype specific OPA titer for at least 1 serotype, or titer/concentration for at least 1 antigen on concomitant vaccines). Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 133 | 122 | 125 | 132
mcg/mL
  Serotype 1 | 1.91 [1.66 to 2.19] | 2.21 [1.88 to 2.61] | 1.97 [1.66 to 2.34] | 2.81 [2.39 to 3.30]
  Serotype 3 | 0.800 [0.721 to 0.887] | 1.14 [1.01 to 1.27] | 1.17 [1.04 to 1.31] | 0.676 [0.598 to 0.764]
  Serotype 4 | 0.900 [0.819 to 0.988] | 0.880 [0.798 to 0.971] | 1.06 [0.951 to 1.18] | 1.63 [1.45 to 1.83]
  Serotype 5 | 3.62 [3.02 to 4.35] | 3.26 [2.70 to 3.95] | 3.00 [2.42 to 3.71] | 1.88 [1.63 to 2.17]
  Serotype 6A | 3.41 [2.93 to 3.96] | 2.77 [2.33 to 3.30] | 3.26 [2.78 to 3.82] | 4.53 [3.93 to 5.21]
  Serotype 6B | 1.95 [1.52 to 2.49] | 1.64 [1.22 to 2.20] | 1.97 [1.51 to 2.59] | 2.87 [2.36 to 3.48]
  Serotype 7F | 3.88 [3.47 to 4.34] | 3.68 [3.27 to 4.14] | 3.45 [3.05 to 3.90] | 3.93 [3.53 to 4.36]
  Serotype 9V | 1.35 [1.18 to 1.55] | 1.16 [0.989 to 1.37] | 1.49 [1.27 to 1.74] | 2.41 [2.12 to 2.74]
  Serotype 14: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 14 | 7.49 [6.36 to 8.81] | 6.83 [5.85 to 7.98] | 6.84 [5.73 to 8.17] | 7.41 [6.20 to 8.86]
  Serotype 18C | 1.67 [1.49 to 1.87] | 1.56 [1.391 to 1.76] | 1.46 [1.31 to 1.63] | 1.92 [1.67 to 2.20]
  Serotype 19A | 1.86 [1.57 to 2.20] | 1.74 [1.43 to 2.11] | 1.86 [1.57 to 2.21] | 2.17 [1.85 to 2.54]
  Serotype 19F: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 19F | 3.32 [2.98 to 3.70] | 3.31 [2.93 to 3.75] | 2.95 [2.51 to 3.46] | 3.70 [3.23 to 4.24]
  Serotype 23F | 2.69 [2.31 to 3.13] | 1.96 [1.69 to 2.28] | 2.05 [1.73 to 2.43] | 1.71 [1.44 to 2.04]
  Serotype 8: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 8 | 3.27 [2.92 to 3.66] | 2.87 [2.55 to 3.22] | 3.08 [2.70 to 3.51] | 0.105 [0.093 to 0.119]
  Serotype 9N | 2.53 [2.26 to 2.84] | 2.39 [2.10 to 2.71] | 2.42 [2.12 to 2.77] | 0.510 [0.424 to 0.612]
  Serotype 10A | 2.86 [2.29 to 3.57] | 2.84 [2.24 to 3.59] | 3.26 [2.68 to 3.97] | 0.098 [0.089 to 0.108]
  Serotype 11A | 2.52 [2.21 to 2.88] | 2.51 [2.21 to 2.85] | 2.32 [1.99 to 2.71] | 0.108 [0.095 to 0.123]
  Serotype 12F | 1.93 [1.68 to 2.23] | 1.56 [1.33 to 1.82] | 1.54 [1.31 to 1.81] | 0.076 [0.075 to 0.078]
  Serotype 15B: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 15B | 7.88 [6.54 to 9.48] | 7.161 [5.73 to 8.95] | 6.84 [5.54 to 8.45] | 0.097 [0.087 to 0.107]
  Serotype 22F | 12.3 [10.8 to 14.1] | 10.4 [8.59 to 12.6] | 9.27 [7.58 to 11.3] | 0.092 [0.083 to 0.103]
  Serotype 33F: number analyzed (Participants) | 133 | 122 | 125 | 131
  Serotype 33F | 2.67 [2.11 to 3.37] | 2.61 [2.05 to 3.32] | 2.57 [2.09 to 3.16] | 0.093 [0.085 to 0.101]

9. Primary Outcome: For Infants: Serotype Specific IgG GMCs for Each Pneumococcal Serotype at 30 Days Post-Dose 4
Description: The GMCs for serotype specific pneumococcal IgG antibodies were measured using PnPS-ECL, a multiplexed serological assay which allows for the simultaneous quantification of human IgG against pneumococcal polysaccharide antigens.
Time Frame: Day 330
Population: Per protocol analysis set 3 (PPAS3) was a subset of Full analysis set 3 (FAS3). FAS3: All randomized participants to Groups 5 to 8 who received at least 1 dose of study vaccine at time of booster and had a valid post-booster vaccination blood sample result (serotype specific IgG concentration or serotype specific OPA titer for at least 1 serotype or titer/concentration for at least 1 antigen on concomitant vaccines). Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 122 | 108 | 101 | 128
mcg/mL
  Serotype 1 | 3.16 [2.68 to 3.73] | 3.59 [3.02 to 4.26] | 3.44 [2.87 to 4.12] | 3.89 [3.35 to 4.50]
  Serotype 3: number analyzed (Participants) | 122 | 108 | 101 | 127
  Serotype 3 | 0.755 [0.675 to 0.844] | 1.07 [0.949 to 1.21] | 1.03 [0.922 to 1.16] | 0.961 [0.843 to 1.09]
  Serotype 4 | 1.37 [1.18 to 1.59] | 1.25 [1.08 to 1.45] | 1.75 [1.49 to 2.05] | 2.41 [2.09 to 2.77]
  Serotype 5 | 7.56 [6.24 to 9.18] | 6.46 [5.25 to 7.95] | 6.63 [5.32 to 8.24] | 3.07 [2.67 to 3.54]
  Serotype 6A | 9.44 [8.01 to 11.1] | 8.08 [6.93 to 9.43] | 7.80 [6.50 to 9.36] | 10.8 [9.36 to 12.4]
  Serotype 6B: number analyzed (Participants) | 122 | 108 | 100 | 128
  Serotype 6B | 8.77 [7.14 to 10.8] | 8.36 [6.88 to 10.2] | 7.96 [6.63 to 9.57] | 8.54 [7.46 to 9.78]
  Serotype 7F | 4.42 [3.93 to 4.97] | 4.19 [3.63 to 4.85] | 3.76 [3.33 to 4.24] | 5.41 [4.80 to 6.09]
  Serotype 9V | 2.20 [1.89 to 2.57] | 2.06 [1.78 to 2.38] | 2.57 [2.20 to 3.01] | 4.32 [3.77 to 4.95]
  Serotype 14 | 6.94 [5.93 to 8.11] | 6.77 [5.62 to 8.14] | 7.70 [6.58 to 9.00] | 8.73 [7.34 to 10.4]
  Serotype 18C | 1.79 [1.58 to 2.02] | 1.66 [1.46 to 1.90] | 1.55 [1.37 to 1.77] | 2.81 [2.46 to 3.21]
  Serotype 19A | 6.92 [5.79 to 8.28] | 7.36 [6.12 to 8.84] | 7.72 [6.37 to 9.36] | 7.38 [6.28 to 8.67]
  Serotype 19F: number analyzed (Participants) | 122 | 108 | 100 | 128
  Serotype 19F | 6.64 [5.75 to 7.67] | 7.48 [6.18 to 9.06] | 6.68 [5.62 to 7.94] | 7.03 [6.05 to 8.16]
  Serotype 23F: number analyzed (Participants) | 122 | 107 | 101 | 128
  Serotype 23F | 3.78 [3.19 to 4.49] | 2.90 [2.46 to 3.42] | 2.99 [2.50 to 3.57] | 3.54 [3.02 to 4.16]
  Serotype 8 | 4.64 [3.94 to 5.46] | 4.36 [3.74 to 5.08] | 4.26 [3.56 to 5.10] | 0.238 [0.196 to 0.289]
  Serotype 9N: number analyzed (Participants) | 121 | 108 | 101 | 128
  Serotype 9N | 4.16 [3.60 to 4.79] | 4.23 [3.72 to 4.80] | 3.80 [3.18 to 4.54] | 0.953 [0.773 to 1.18]
  Serotype 10A | 5.67 [4.71 to 6.83] | 5.70 [4.76 to 6.83] | 4.78 [3.96 to 5.78] | 0.160 [0.137 to 0.187]
  Serotype 11A | 3.66 [3.17 to 4.21] | 3.92 [3.36 to 4.57] | 3.22 [2.69 to 3.85] | 0.154 [0.128 to 0.186]
  Serotype 12F | 2.68 [2.30 to 3.13] | 2.25 [1.94 to 2.61] | 2.04 [1.73 to 2.41] | 0.080 [0.076 to 0.085]
  Serotype 15B: number analyzed (Participants) | 122 | 108 | 101 | 126
  Serotype 15B | 19.6 [16.5 to 23.2] | 17.3 [14.2 to 21.2] | 15.7 [12.6 to 19.5] | 0.114 [0.097 to 0.134]
  Serotype 22F: number analyzed (Participants) | 122 | 108 | 100 | 128
  Serotype 22F | 24.5 [21.1 to 28.3] | 21.3 [17.8 to 25.6] | 20.6 [16.8 to 25.2] | 0.173 [0.144 to 0.206]
  Serotype 33F | 4.74 [4.07 to 5.52] | 4.83 [4.13 to 5.65] | 4.62 [3.89 to 5.49] | 0.158 [0.134 to 0.186]

10. Secondary Outcome: For Toddlers: Serotype Specific OPA Geometric Mean Titers (GMTs) for Each Pneumococcal Serotype 30 Days Post-Dose
Description: The GMs for serotype specific OPA titers were measured using multiplex opsonophagocytic assay (MOPA) which is used to evaluate the opsonophagocytic index (50% killing) of pneumococcal anti-capsular polysaccharide antibodies in human serum samples following vaccination.
Time Frame: Day 30
Population: Results are based on PPAS1 which is a subset of the FAS1 for toddlers. Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution (1/dil)
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13
Number analyzed (Participants) | 24 | 24 | 23 | 25
1/dilution (1/dil)
  Serotype 1 | 138 [62.1 to 306] | 94.2 [49.9 to 178] | 177 [92.3 to 339] | 247 [140 to 434]
  Serotype 3: number analyzed (Participants) | 24 | 22 | 22 | 25
  Serotype 3 | 272 [204 to 363] | 314 [229 to 431] | 393 [287 to 537] | 216 [160 to 292]
  Serotype 4: number analyzed (Participants) | 24 | 23 | 23 | 25
  Serotype 4 | 3467 [2296 to 5234] | 2862 [2027 to 4041] | 5420 [3366 to 8725] | 2975 [1981 to 4466]
  Serotype 5: number analyzed (Participants) | 24 | 23 | 22 | 25
  Serotype 5 | 1287 [736 to 2252] | 1333 [867 to 2050] | 1397 [817 to 2389] | 1307 [820 to 2082]
  Serotype 6A: number analyzed (Participants) | 24 | 21 | 22 | 25
  Serotype 6A | 4623 [3110 to 6871] | 6083 [4341 to 8523] | 7232 [5071 to 10315] | 7553 [5386 to 10592]
  Serotype 6B: number analyzed (Participants) | 24 | 23 | 23 | 25
  Serotype 6B | 3027 [1935 to 4737] | 3542 [2348 to 5342] | 5171 [3369 to 7935] | 4679 [3132 to 6992]
  Serotype 7F | 8449 [5127 to 13924] | 7640 [4974 to 11734] | 6284 [4099 to 9634] | 10443 [6580 to 16575]
  Serotype 9V: number analyzed (Participants) | 24 | 22 | 22 | 24
  Serotype 9V | 3612 [2492 to 5236] | 3254 [2121 to 4991] | 4720 [2911 to 7654] | 4057 [2778 to 5926]
  Serotype 14: number analyzed (Participants) | 24 | 24 | 22 | 25
  Serotype 14 | 3598 [2195 to 5898] | 3881 [2534 to 5943] | 3191 [2045 to 4979] | 2828 [1948 to 4107]
  Serotype 18C: number analyzed (Participants) | 24 | 22 | 23 | 25
  Serotype 18C | 1490 [921 to 2411] | 1760 [1176 to 2634] | 1722 [1233 to 2404] | 2424 [1558 to 3771]
  Serotype 19A: number analyzed (Participants) | 24 | 22 | 23 | 24
  Serotype 19A | 3082 [2115 to 4493] | 3174 [2302 to 4377] | 3004 [2121 to 4256] | 5354 [3343 to 8577]
  Serotype 19F: number analyzed (Participants) | 24 | 23 | 22 | 25
  Serotype 19F | 1194 [838 to 1701] | 1806 [1207 to 2702] | 1569 [955 to 2576] | 2554 [1818 to 3588]
  Serotype 23F: number analyzed (Participants) | 24 | 23 | 22 | 25
  Serotype 23F | 5451 [3431 to 8662] | 7457 [5131 to 10838] | 5179 [3303 to 8121] | 9264 [5738 to 14957]
  Serotype 8: number analyzed (Participants) | 24 | 23 | 23 | 25
  Serotype 8 | 4244 [2705 to 6658] | 7003 [5065 to 9681] | 7989 [5076 to 12576] | 222 [120 to 412]
  Serotype 9N: number analyzed (Participants) | 24 | 23 | 23 | 25
  Serotype 9N | 11562 [9510 to 14057] | 8391 [6117 to 11511] | 12115 [8129 to 18054] | 2061 [1445 to 2940]
  Serotype 10A: number analyzed (Participants) | 24 | 23 | 23 | 24
  Serotype 10A | 3582 [2518 to 5096] | 3615 [2706 to 4829] | 4001 [2768 to 5782] | 10.0 [4.07 to 24.7]
  Serotype 11A: number analyzed (Participants) | 24 | 24 | 23 | 24
  Serotype 11A | 611 [378 to 988] | 686 [349 to 1345] | 661 [311 to 1408] | 4.14 [3.86 to 4.44]
  Serotype 12F: number analyzed (Participants) | 24 | 21 | 21 | 25
  Serotype 12F | 6767 [4628 to 9895] | 7391 [4704 to 11615] | 7955 [4793 to 13205] | 5.27 [3.28 to 8.46]
  Serotype 15B: number analyzed (Participants) | 21 | 19 | 21 | 24
  Serotype 15B | 1087 [402 to 2941] | 1346 [496 to 3658] | 1476 [467 to 4671] | 37.7 [20.3 to 69.8]
  Serotype 22F: number analyzed (Participants) | 22 | 24 | 22 | 25
  Serotype 22F | 4106 [2963 to 5690] | 3352 [2354 to 4773] | 4443 [2858 to 6906] | 69.0 [24.3 to 196]
  Serotype 33F | 39691 [27999 to 56266] | 30399 [18394 to 50238] | 35326 [24106 to 51770] | 2689 [1702 to 4249]

11. Secondary Outcome: For Infants: Serotype Specific OPA GMTs for Each Pneumococcal Serotype 30 Days Post-Dose 3
Description: The GMs for serotype specific OPA titers were measured using MOPA which is used to evaluate the opsonophagocytic index (50% killing) of pneumococcal anti-capsular polysaccharide antibodies in human serum samples following vaccination.
Time Frame: Day 150
Population: Results are based on PPPAS2-OPA subset which is a subset of the FAS for infants. Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dil
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 89 | 85 | 83 | 95
1/dil
  Serotype 1 | 73.6 [53.4 to 101] | 81.7 [59.1 to 113] | 66.4 [46.7 to 94.5] | 114 [86.4 to 151]
  Serotype 3: number analyzed (Participants) | 89 | 85 | 82 | 93
  Serotype 3 | 170 [146 to 197] | 218 [180 to 266] | 260 [226 to 300] | 178 [147 to 215]
  Serotype 4: number analyzed (Participants) | 87 | 85 | 83 | 95
  Serotype 4 | 703 [586 to 843] | 616 [492 to 771] | 1154 [934 to 1425] | 1789 [1489 to 2151]
  Serotype 5 | 602 [469 to 771] | 492 [372 to 652] | 495 [370 to 662] | 569 [450 to 719]
  Serotype 6A | 2456 [2032 to 2969] | 2223 [1743 to 2834] | 2664 [2187 to 3245] | 2799 [2307 to 3395]
  Serotype 6B | 1436 [1008 to 2045] | 1041 [677 to 1602] | 1885 [1384 to 2567] | 2472 [1934 to 3160]
  Serotype 7F | 5964 [4989 to 7130] | 5449 [4536 to 6545] | 5889 [4980 to 6963] | 5252 [4521 to 6102]
  Serotype 9V: number analyzed (Participants) | 89 | 85 | 81 | 95
  Serotype 9V | 898 [659 to 1224] | 700 [483 to 1014] | 1136 [866 to 1492] | 1319 [1040 to 1672]
  Serotype 14 | 1959 [1580 to 2429] | 1767 [1391 to 2244] | 2293 [1858 to 2829] | 1920 [1574 to 2344]
  Serotype 18C | 866 [731 to 1026] | 819 [668 to 1003] | 804 [660 to 979] | 1000 [804 to 1245]
  Serotype 19A | 640 [521 to 788] | 512 [384 to 684] | 778 [630 to 962] | 1130 [959 to 1332]
  Serotype 19F | 533 [422 to 674] | 591 [451 to 774] | 629 [461 to 860] | 613 [489 to 768]
  Serotype 23F: number analyzed (Participants) | 89 | 85 | 83 | 93
  Serotype 23F | 2654 [2157 to 3265] | 1967 [1500 to 2580] | 2279 [1770 to 2934] | 4299 [3536 to 5227]
  Serotype 8 | 1486 [1239 to 1782] | 1440 [1237 to 1677] | 1612 [1378 to 1886] | 133 [89.9 to 196]
  Serotype 9N: number analyzed (Participants) | 89 | 85 | 83 | 94
  Serotype 9N | 4261 [3534 to 5138] | 4994 [4248 to 5870] | 5257 [4150 to 6661] | 811 [585 to 1126]
  Serotype 10A: number analyzed (Participants) | 89 | 85 | 83 | 94
  Serotype 10A | 2306 [1539 to 3453] | 2722 [1875 to 3951] | 3251 [2501 to 4225] | 9.42 [6.33 to 14.0]
  Serotype 11A: number analyzed (Participants) | 88 | 85 | 81 | 94
  Serotype 11A | 52.6 [36.7 to 75.3] | 64.9 [44.2 to 95.3] | 76.6 [52.6 to 112] | 5.91 [4.62 to 7.54]
  Serotype 12F: number analyzed (Participants) | 89 | 85 | 83 | 94
  Serotype 12F | 2182 [1764 to 2700] | 2179 [1798 to 2640] | 2334 [1836 to 2967] | 5.31 [4.15 to 6.80]
  Serotype 15B: number analyzed (Participants) | 86 | 85 | 81 | 93
  Serotype 15B | 6686 [5281 to 8466] | 5859 [4218 to 8139] | 5220 [3829 to 7116] | 28.1 [22.8 to 34.7]
  Serotype 22F | 5227 [4421 to 6181] | 4657 [3802 to 5706] | 4617 [3725 to 5723] | 16.1 [12.5 to 20.7]
  Serotype 33F: number analyzed (Participants) | 89 | 83 | 83 | 90
  Serotype 33F | 10070 [7198 to 14088] | 11179 [8604 to 14524] | 11900 [8552 to 16559] | 311 [181 to 535]

12. Secondary Outcome: For Infants: Serotype Specific OPA GMTs for Each Pneumococcal Serotype 30 Days Post-Dose 4
Description: as for outcome 11
Time Frame: Day 330
Population: Results are based on PPAS3-OPA subset which is a subset of the FAS3 for infants. Only participants with data collected for each specified category are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dil
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 82 | 73 | 70 | 92
1/dil
  Serotype 1: number analyzed (Participants) | 82 | 73 | 69 | 92
  Serotype 1 | 407 [295 to 561] | 355 [255 to 495] | 320 [211 to 486] | 318 [251 to 403]
  Serotype 3: number analyzed (Participants) | 82 | 70 | 69 | 87
  Serotype 3 | 274 [230 to 328] | 308 [244 to 390] | 376 [314 to 450] | 348 [294 to 412]
  Serotype 4: number analyzed (Participants) | 81 | 72 | 70 | 85
  Serotype 4 | 3754 [3002 to 4694] | 2536 [1915 to 3359] | 5556 [4318 to 7150] | 6028 [4801 to 7570]
  Serotype 5: number analyzed (Participants) | 82 | 72 | 68 | 92
  Serotype 5 | 2348 [1884 to 2926] | 1787 [1365 to 2339] | 2131 [1626 to 2794] | 1396 [1119 to 1740]
  Serotype 6A: number analyzed (Participants) | 82 | 72 | 69 | 90
  Serotype 6A | 5153 [4338 to 6119] | 4786 [3929 to 5829] | 4433 [3434 to 5722] | 6862 [5741 to 8202]
  Serotype 6B: number analyzed (Participants) | 81 | 72 | 70 | 91
  Serotype 6B | 3899 [3019 to 5037] | 3305 [2614 to 4178] | 3638 [2756 to 4802] | 7092 [5699 to 8825]
  Serotype 7F: number analyzed (Participants) | 82 | 72 | 69 | 90
  Serotype 7F | 10234 [8469 to 12368] | 8643 [7263 to 10285] | 9232 [7448 to 11444] | 13971 [11575 to 16863]
  Serotype 9V: number analyzed (Participants) | 80 | 71 | 69 | 86
  Serotype 9V | 3044 [2424 to 3823] | 2641 [2137 to 3263] | 2956 [2363 to 3698] | 4364 [3459 to 5505]
  Serotype 14 | 3415 [2785 to 4188] | 3098 [2527 to 3798] | 4190 [3397 to 5168] | 3378 [2559 to 4459]
  Serotype 18C: number analyzed (Participants) | 82 | 72 | 68 | 92
  Serotype 18C | 1891 [1565 to 2285] | 1422 [1110 to 1823] | 1368 [1092 to 1713] | 2821 [2342 to 3399]
  Serotype 19A: number analyzed (Participants) | 80 | 70 | 67 | 82
  Serotype 19A | 3808 [3057 to 4743] | 3086 [2422 to 3933] | 3580 [2806 to 4566] | 7535 [6068 to 9357]
  Serotype 19F: number analyzed (Participants) | 81 | 71 | 69 | 88
  Serotype 19F | 2071 [1730 to 2481] | 1821 [1313 to 2527] | 1654 [1173 to 2332] | 2249 [1750 to 2889]
  Serotype 23F: number analyzed (Participants) | 80 | 71 | 67 | 87
  Serotype 23F | 5444 [4211 to 7037] | 4444 [3644 to 5418] | 4047 [3019 to 5424] | 18569 [14765 to 23352]
  Serotype 8 | 4559 [3753 to 5537] | 4229 [3527 to 5070] | 4916 [3751 to 6443] | 773 [616 to 970]
  Serotype 9N: number analyzed (Participants) | 81 | 71 | 70 | 90
  Serotype 9N | 9479 [7967 to 11277] | 8565 [7485 to 9800] | 10257 [8771 to 11995] | 3043 [2370 to 3906]
  Serotype 10A: number analyzed (Participants) | 82 | 73 | 70 | 81
  Serotype 10A | 4278 [3125 to 5856] | 4797 [3722 to 6184] | 4768 [3358 to 6770] | 46.6 [23.9 to 90.9]
  Serotype 11A: number analyzed (Participants) | 82 | 73 | 66 | 85
  Serotype 11A | 433 [310 to 604] | 390 [253 to 603] | 550 [372 to 812] | 8.11 [5.45 to 12.1]
  Serotype 12F: number analyzed (Participants) | 81 | 69 | 69 | 75
  Serotype 12F | 4520 [3743 to 5459] | 4757 [3800 to 5956] | 5030 [3785 to 6685] | 7.92 [5.26 to 12.0]
  Serotype 15B: number analyzed (Participants) | 78 | 72 | 67 | 82
  Serotype 15B | 14756 [11612 to 18750] | 13136 [9623 to 17932] | 12799 [9111 to 17981] | 55.2 [36.7 to 83.0]
  Serotype 22F: number analyzed (Participants) | 79 | 71 | 63 | 80
  Serotype 22F | 20372 [15640 to 26536] | 16063 [12306 to 20967] | 21319 [15648 to 29045] | 65.7 [37.7 to 114]
  Serotype 33F: number analyzed (Participants) | 81 | 70 | 66 | 90
  Serotype 33F | 26134 [20845 to 32766] | 21202 [17071 to 26332] | 32376 [25782 to 40657] | 3224 [2388 to 4353]

13. Secondary Outcome: For Infants: GMC of Anti-Rotavirus Serum Immunoglobulin A (IgA) Antibodies 30 Days Post-Dose 3
Description: Anti-rotavirus IgA antibodies in human serum were measured by enzyme linked immunosorbent assay (ELISA). A reference standard assayed on each plate was used to calculate the amount of specific anti-rotavirus IgA antibody in the units assigned by the reference standard.
Time Frame: Day 150
Population: Results are based on PPAS2 which is a subset of the FAS2 for infants. Only participants with data collected for this outcome measure are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Units (U)/mL
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 119 | 105 | 110 | 120
Units (U)/mL | 407 [303 to 545] | 390 [283 to 537] | 494 [369 to 661] | 393 [277 to 560]

14. Secondary Outcome: For Infants: Percentage of Participants With Antibody Responses to Diphtheria, Tetanus and Polyribosylribitol Phosphate Antigens 30 Days Post-Dose 3
Description: Percentage of participants with toxoid concentration >=0.10 mcg/mL for diphtheria and tetanus and >=0.15 mcg/mL for PRP are presented. Anti-diphtheria and anti-tetanus concentrations were measured using electro-chemiluminescence assay (ECL) and anti-PRP concentrations were measured using a Farr-type radioimmunoassay.
Time Frame: Day 150
Population: Results are based on PPAS2 which is a subset of the FAS2 for infants. Only participants with data collected for each specified category are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 130 | 118 | 123 | 130
percentage of participants
  Anti-Diphtheria toxoid | 94.6 [89.2 to 97.8] | 97.5 [92.7 to 99.5] | 95.9 [90.8 to 98.7] | 96.9 [92.3 to 99.2]
  Anti-Tetanus toxoid | 100 [97.2 to 100] | 100 [96.9 to 100] | 100 [97.0 to 100] | 100 [97.2 to 100]
  Anti-PRP: number analyzed (Participants) | 127 | 113 | 112 | 128
  Anti-PRP | 99.2 [95.7 to 100] | 99.1 [95.2 to 100] | 98.2 [93.7 to 99.8] | 100 [97.2 to 100]

15. Secondary Outcome: For Infants: Percentage of Participants With Antibody Responses to Poliovirus 1, 2 and 3 30 Days Post-Dose 3
Description: Anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. Response was defined as a titer >=8.
Time Frame: Day 150
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 125 | 109 | 114 | 127
percentage of participants
  Anti-poliovirus 1: number analyzed (Participants) | 123 | 109 | 114 | 126
  Anti-poliovirus 1 | 99.2 [95.6 to 100] | 100 [96.7 to 100] | 97.4 [92.5 to 99.5] | 100 [97.1 to 100]
  Anti-poliovirus 2: number analyzed (Participants) | 122 | 105 | 112 | 124
  Anti-poliovirus 2 | 100 [97.0 to 100] | 100 [96.5 to 100] | 99.1 [95.1 to 100] | 100 [97.1 to 100]
  Anti-poliovirus 3: number analyzed (Participants) | 125 | 109 | 111 | 127
  Anti-poliovirus 3 | 100 [97.1 to 100] | 100 [96.7 to 100] | 99.1 [95.1 to 100] | 100 [97.1 to 100]

16. Secondary Outcome: For Infants: GMCs of Antibodies to Pertussis Antigens 30 Days Post-Dose 3
Description: Serum samples were collected for analysis by ECL to determine the GMC of antibodies to the following Pertussis antigens: Pertussis toxoid/toxin, Filamentous hemagglutinin, Pertactin and Fimbriae types 2 and 3.
Time Frame: Day 150
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units (EU)/mL
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 130 | 118 | 123 | 130
ELISA units (EU)/mL
  Pertussis toxoid/toxin | 67.9 [60.1 to 76.6] | 77.2 [67.4 to 88.5] | 66.3 [57.4 to 76.6] | 68.3 [59.7 to 78.2]
  Filamentous hemagglutinin | 109 [94.9 to 124] | 107 [94.4 to 122] | 108 [95.2 to 123] | 104 [93.0 to 116]
  Pertactin | 38.3 [32.3 to 45.4] | 36.1 [29.4 to 44.3] | 39.8 [32.8 to 48.3] | 45.2 [37.7 to 54.1]
  Fimbriae types 2 and 3 | 347 [295 to 408] | 341 [286 to 407] | 315 [262 to 380] | 343 [282 to 418]

17. Secondary Outcome: For Infants: Percentage of Participants With Antibody Responses to Hepatitis-B Antigens 30 Days Post-Dose 3
Description: Anti-Hepatitis B antibodies were measured by the commercially available VITROS ECi/ECiQ immunodiagnostic system using chemiluminescence detection technology. The VITROS ECi immunodiagnostic system uses an antibody mediated antigen sandwich formation to detect the presence of anti-hepatitis B surface antigen total immunoglobulin in human serum. The threshold presented is >=10 milli international units (mIU).
Time Frame: Day 150
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 121 | 106 | 108 | 123
percentage of participants | 98.3 [94.2 to 99.8] | 99.1 [94.9 to 100] | 98.1 [93.5 to 99.8] | 99.2 [95.6 to 100]

18. Secondary Outcome: For Infants: Percentage of Participants With Antibody Responses to M-MRII and Varivax Antigens 30 Days Post-Dose 4
Description: Anti-measles antibodies were determined by bulk measles IgG enzyme immunoassay (EIA); anti-mumps antibodies by ELISA, anti-rubella antibodies by bulk rubella IgG EIA and anti-varicella antibodies were determined by glycoprotein ELISA to detect total IgG antibody to respective virus before and after vaccination with a virus-containing vaccine. Percentage of participants with anti-measles antibody concentrations >=255 mIU/mL, anti-mumps antibody concentrations: >=10 antibody units/mL, anti-rubella antibody concentrations >=10 IU/mL and anti-varicella concentrations >=5 units/mL is reported in this outcome measure.
Time Frame: Day 330
Population: Results are based on PPAS3 which is a subset of the FAS3 for infants. Only participants with data collected for this outcome measure are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
Number analyzed (Participants) | 118 | 104 | 98 | 124
percentage of participants
  Anti-Measles | 97.5 [92.7 to 99.5] | 97.1 [91.8 to 99.4] | 96.9 [91.3 to 99.4] | 98.4 [94.3 to 99.8]
  Anti-Mumps | 99.2 [95.4 to 100] | 97.1 [91.8 to 99.4] | 96.9 [91.3 to 99.4] | 98.4 [94.3 to 99.8]
  Anti-Rubella | 98.3 [94.0 to 99.8] | 98.1 [93.2 to 99.8] | 99.0 [94.4 to 100] | 98.4 [94.3 to 99.8]
  Anti-Varicella | 100 [96.9 to 100] | 99.0 [94.8 to 100] | 95.9 [89.9 to 98.9] | 98.4 [94.3 to 99.8]

ADVERSE EVENTS:
Time Frame: AEs data was collected from first dose vaccine administration (Day 1) until 6 months after the last dose administration, 490 days. All-cause mortality was collected up to end of the study (Stage I: 6 months and Stage II: 19 months)
Description: Analysis was performed on the safety analysis set. One participant who was randomized to the reporting group "Stage II: Group 7 SP0202-VII" was administered SP0202-IIb formulation. Therefore, the participant was included in "Stage II: Group 5 SP0202-IIb" for analysis.
Arm/Group | Stage I: Group 1 SP0202-IIb | Stage I: Group 2 SP0202-VI | Stage I: Group 3 SP0202-VII | Stage I: Group 4 Prevnar 13 | Stage II: Group 5 SP0202-IIb | Stage II: Group 6 SP0202-VI | Stage II: Group 7 SP0202-VII | Stage II: Group 8 Prevnar 13
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34 | 0/35 | 0/34 | 0/180 | 1/178 | 0/176 | 0/176
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/34 | 0/35 | 0/34 | 3/180 | 9/178 | 8/176 | 9/176
Other Adverse Events (participants affected / at risk) | 28/35 | 28/34 | 29/35 | 25/34 | 160/180 | 164/178 | 159/176 | 158/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I: Group 1 SP0202-IIb (N=35) | Stage I: Group 2 SP0202-VI (N=34) | Stage I: Group 3 SP0202-VII (N=35) | Stage I: Group 4 Prevnar 13 (N=34) | Stage II: Group 5 SP0202-IIb (N=180) | Stage II: Group 6 SP0202-VI (N=178) | Stage II: Group 7 SP0202-VII (N=176) | Stage II: Group 8 Prevnar 13 (N=176)
Heart Disease Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial Diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb Asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I: Group 1 SP0202-IIb (N=35) | Stage I: Group 2 SP0202-VI (N=34) | Stage I: Group 3 SP0202-VII (N=35) | Stage I: Group 4 Prevnar 13 (N=34) | Stage II: Group 5 SP0202-IIb (N=180) | Stage II: Group 6 SP0202-VI (N=178) | Stage II: Group 7 SP0202-VII (N=176) | Stage II: Group 8 Prevnar 13 (N=176)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 18 (22) | 16 (18) | 17 (20) | 25 (26)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 43 (65) | 36 (58) | 43 (60) | 45 (58)
Crying (General disorders) | 16 (16) | 6 (6) | 17 (17) | 17 (17) | 113 (230) | 112 (224) | 101 (204) | 106 (231)
Injection Site Bruising (General disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 11 (17) | 10 (14) | 14 (29) | 17 (23)
Injection Site Erythema (General disorders) | 20 (31) | 14 (25) | 13 (21) | 10 (18) | 71 (269) | 58 (213) | 65 (282) | 65 (260)
Injection Site Pain (General disorders) | 16 (26) | 12 (20) | 19 (34) | 13 (23) | 120 (673) | 127 (757) | 125 (736) | 124 (816)
Injection Site Swelling (General disorders) | 16 (24) | 14 (21) | 14 (22) | 9 (16) | 50 (186) | 48 (171) | 49 (166) | 59 (203)
Pyrexia (General disorders) | 4 (4) | 7 (7) | 8 (8) | 9 (9) | 67 (108) | 61 (82) | 63 (90) | 68 (97)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 11 (12) | 8 (10) | 8 (8)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 61 (92) | 55 (78) | 61 (92) | 48 (73)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 4 (5) | 4 (4) | 10 (11)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 10 (11) | 6 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 8 (8) | 5 (5) | 10 (12)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9) | 7 (7) | 13 (13) | 11 (11) | 70 (118) | 70 (109) | 68 (110) | 67 (118)
Somnolence (Nervous system disorders) | 12 (12) | 11 (11) | 12 (12) | 10 (10) | 94 (209) | 97 (211) | 92 (209) | 104 (220)
Irritability (Psychiatric disorders) | 21 (21) | 16 (16) | 22 (22) | 20 (20) | 110 (270) | 116 (278) | 114 (262) | 117 (289)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04398706/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT04398706/SAP_001.pdf